CLINICAL TRIAL: NCT00797329
Title: Biological and Cognitive Markers of Violent Behavior in Forensic Patients With Polysubstance Use: Retrospective Evaluation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: BeerYaakov Mental Health Center (Other Government)
Responsible Party: Dr. Kertzman, BeerYaakov Mental Health Center
Other Study IDs: 222CTIL
Record Dates: First submitted 2008-11-23; First posted 2008-11-25 (Estimated); Last update posted 2008-11-25 (Estimated); Status verified 2008-11

CONDITIONS: Violent Behavior; Polydrug Use; Alcohol Abuse
Keywords: psychiatric patients with violent behavior
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Time Perspective: Retrospective

GROUPS / COHORTS (1):
- observation: adult men with alcohol and polydrug use according to DSM-IV criteria, hospitalized in maximum security department between 2002 - 2008
  Interventions: Other: chart review

INTERVENTIONS:
Other: chart review — * cholesterol
  * cognitive profiles
  * violent behavior

SUMMARY:
Aggressive behavior, both in the form of violence toward others (injury-inflicting or homicide) or toward oneself (suicide or self-injures) create problems of patient management, treatment and paroles.

Biological causes of violent crime were hypothesized by Eysenck (1978), who believed that criminality resulted from a nervous system distinct from that of most people.

The prefrontal cortex, regulates planning of motor acts and executive functions, which are critical for inhibitory ability and control of impulsive outburst were found to be impaired in violent subjects (Hoaken et al, 2003; Blair, 2001; Brower and Price, 2001; Filley et al, 2001; Raine et al, 2000; George et al, 2004; Dolan and Park, 2002; Stevens et al, 2003; Raine and Yang, 2006), especially in impulsive offenders murderers (Raine et al, 1997; 1998). Violence act influenced by nonplaning outboards definite as impulsive aggression (Linnoila and Charney, 1999), which one of the most important factor influenced by dangerous behavior in general (for review: Skodol, 1998, Moeller et al, 2001; Pontius, 2000; 2004; Siever, 2008).

Cholesterol and fats have many roles and may influence brain function and behavior through modification of membranes; myelin; enzyme function; absorption and transport of fat-soluble vitamins and toxins; and steroid hormones and through effects on production, reuptake, or metabolism of neurotransmitters (Boston et al, 1996).

Since 80-th a strong association was found between low cholesterol levels and violent behavior, an association that was not due to age, race, sex, or diagnosis (Mufti et al, 1998; New et al, 1999; Alvarez et al, 2000; Golomb et al, 2000; Hillbrand et al, 2000; Troisi and D'Argenio, 2006; Chakrabarat and Sinha, 2006).

Associations between violent behavior, cognitive functioning and total cholesterol level were contradicted with difference in samples and behavioral parameters: homicide, homicide attempts, rape, physical or verbal aggression, complete suicide or suicide attempts, only partially accounted for each measure of behaviors, suggesting that further investigation is warranted. Because of the inconsistencies in the available data, we studied retrospectively a group of criminal offenders with alcohol and drug use. Our analysis of lipid constituents in serum focused on TC, HDL, LDL, and TG.

Significance of the study. It is possible that cholesterol profile is a biomarker and potential predictor of violent in patients with polydrug use.

The purpose of this retrospective study is to investigate the correlations between cholesterol and cognitive profiles in psychiatric patients with violent behaviour. The demographic and criminal records, clinical characteristics, cholesterol profiles, and cognitive performance data of these patients will be will be intercorrelated.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 19-65 years
2. Men with verified diagnoses of alcohol and polydrug use according to DSM-IV criteria, underwent cholesterol and cognitive assessment, while being incarcerated in maximum-security forensic facility

Exclusion Criteria:

1. Subjects suffering from any clinically significant metabolic disorder (e.g. diabetes, hypo-hyperthiorioidosis, et ctr)
2. Subjects suffering from clinically significant infectional disorder (e.g. tuberculosis, pneumonia, AIDS, active HCV et ctr)
3. Subjects starving or suffering from severe hepatic or kidney dysfunction and insufficiency
4. patients with comorbid diagnoses of schizophrenia, schizoaffective disorder and bipolar mood disorder
5. patients with comorbide mild mental retardation or epilepsy
6. patients with using cholesterol lowering agent

Ages: 19 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age between 19-65 years; men with verified diagnoses of alcohol and polydrug use according to DSM-IV criteria; hospitalized in maximum security department between 2002 - 2008.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-07

PRIMARY OUTCOMES:
The purpose of this retrospective study is to investigate the correlations between cholesterol and cognitive profiles in psychiatric patients with violent behaviour. | 2008-2009

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Beer-Yaacov MHC, Beer Yaacov
  - BeerYaakov MHC, Beer Yaakov